CLINICAL TRIAL: NCT05490901
Title: A Retrospective and Prospective Cohort Study to Investigate the Prognostic Role and Diagnostic Efficacy of Exercise Right Heart Catheterization With a Simultaneous Echocardiography in Patients With Dyspnea on Exertion
Brief Title: The Prognostic Role and Diagnostic Efficacy of Exercise Right Heart Catheterization With a Simultaneous Echocardiography in Patients With Dyspnea on Exertion
Acronym: EX_CATH
Status: Recruiting | Type: Observational
Sponsor: Samsung Medical Center (Other)
Responsible Party: Principal Investigator, Jeong Hoon Yang, Professor, Samsung Medical Center
Other Study IDs: EX_CATH
Record Dates: First submitted 2022-08-01; First posted 2022-08-08 (Actual); Last update posted 2022-08-08 (Actual); Status verified 2022-08

CONDITIONS: Heart Failure With Preserved Ejection Fraction; Chronic Pulmonary Thromboembolism (Disorder)
Keywords: Exercise hemodynamic test; Heart failure with preserved ejection fraction; Cardiac catheterization

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with Unexplained Dyspnea: Patients with dyspnea on exertion
  Interventions: Diagnostic Test: Exercise hemodynamic test

INTERVENTIONS:
Diagnostic Test: Exercise hemodynamic test — Assessment of pulmonary hemodynamics during exercise by right heart catheterization and cardiac function during exercise by a simultaneous transthoracic echocardiography
  Other Names: Exercise cath

SUMMARY:
To evaluate the role of exercise hemodynamic testing in the diagnostic workup for patients with dyspnea on exertion referred to the catheterization lab.

DETAILED DESCRIPTION:
Heart failure with preserved ejection fraction (HFpEF) is a major public health problem that has no proven effective treatment. However, in practice, it's difficult to recognize early stage of HFpEF by resting hemodynamic study and echocardiography because the patients mainly complaint of dyspnea only during exercise but not resting condition. Accordingly, exercise stress test will be helpful to provide more information on pathophysiology, diagnosis, and severity in various cardiovascular diseases such as HFpEF, valvular heart disease, and chronic thromboembolic pulmonary hypertension. Thus, the broad objective of this proposal is to characterize the dynamic changes in cardiopulmonary mechanics during stress in patients with exertional dyspnea, establishing a comprehensive multimodality diagnostic approach to the evaluation of exercise intolerance. Specifically, this study will compare established and novel parameters derived from echocardiography and CPX with simultaneous, gold standard invasive measures of cardiovascular hemodynamics at rest and with exercise stress to define the role of noninvasive testing in the diagnostic workup for patients with dyspnea on exertion referred to the catheterization lab.

ELIGIBILITY:
Inclusion Criteria:

* Subject must be at least 19 years of age.
* Patients with dyspnea on exertion
* Written informed consent of participating subjects after being fully briefed (for prospective analysis)

Exclusion Criteria:

* Patients with incomplete hemodynamic data at rest or exercise
* Advanced tumor disease or other diseases with a short life expectancy
* Uncontrolled systemic arterial hypertension ( > 160/100 mmHg at rest)
* FEV1<50% predicted
* TLC<60% predicted

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients with dyspnea on exertion who undergo right heart catheterization and echocardiography during exercise due to clinical reasons.
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2020-03-17 (Actual); Primary Completion 2028-12-31 (Estimated); Study Completion 2029-06-30 (Estimated)

PRIMARY OUTCOMES:
Proportion of exercise induced pulmonary artery wedge pressure >25 mmHg | during the procedure
  Number of Participants with Diagnosis of earlier heart failure with preserved ejection fraction based on exercise PCWP

SECONDARY OUTCOMES:
Proportion of exercise induced pulmonary hypertension > 30 mmHg | during the procedure
  Number of Participants with Diagnosis of pulmonary hypertension based on mean pulmonary pressure at peak exercise
Correlation between peripheral venous pressure and right atrial pressure assumed by echocardiography | during the procedure
  Correlation between peripheral venous pressure and right atrial pressure assumed by echocardiography
Ventilatory mechanics | during the procedure
  ratio of minute ventilation to carbon dioxide production (VE/VCO2)
Aerobic capacity | during the procedure
  peak oxygen consumption (VO2)
coronary flow reserve | during the procedure
  invasively measured coronary flow reserve
index of microcirculatory resistance | during the procedure
  invasively measured index of microcirculatory resistance
Lactate level at peak exercise | during the procedure
  Serum lactate level at peak exercise
LA stiffness | during the procedure
  LA stiffness measured by LA strain/E/e' using Transthoracic echocardiography
change of E/e' between at rest and peak exercise | between at rest and peak exercise
  The change of E/e' between at rest and peak exercise
Rates of rehospitalization due to heart failure | 5 years follow-up
  Rehospitalization due to heart failure
Rates of all-cause death | 5 years follow-up
  Follow-up death
The change of right ventricular systolic pressure (RVSP) between at rest and peak exercise | between at rest and peak exercise
  The change of RVSP between at rest and peak exercise
change of Tricuspid annular plane systolic excursion (TAPSE) between at rest and peak exercise | between at rest and peak exercise
  The change of TAPSE between at rest and peak exercise
change of S' between at rest and peak exercise | between at rest and peak exercise
  The change of S' between at rest and peak exercise

CONTACTS AND LOCATIONS:
Overall Officials: Jeong Hoon Yang, MD, Principal Investigator — Samsung Medical Center
Locations (1):
- Samsung Medical Center, Seoul, South Korea